CLINICAL TRIAL: NCT02549196
Title: A Phase II, Dose Titration Study of CPC-201 in Patients With Dementia of Alzheimer's Type
Brief Title: A Dose Titration Study of CPC-201 in Patients With Dementia of Alzheimer's Type
Acronym: CPC-12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chase Pharmaceuticals Corporation, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CPC-001-12
Record Dates: First submitted 2015-08-27; First posted 2015-09-15 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Dementia of Alzheimer's Type
MeSH Terms: interventions — Donepezil; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Donepezil 20mg/day upward dose titration of 10mg at weekly intervals up to first intolerable dose (FID) or to maximum allowed dose (MAD) of 60mg/day with solifenacin 15 or 20mg/day.
  Interventions: Drug: Donepezil; Drug: Solifenacin
- Cohort 2 (Experimental): Donepezil 20mg/day upward dose titration of 20mg at weekly intervals up to first intolerable dose (FID) or to maximum allowed dose (MAD) of 60mg/day with solifenacin 15 or 20mg/day.
  Interventions: Drug: Donepezil; Drug: Solifenacin
- Cohort 1b (Experimental): Donepezil 10mg/day upward dose titration of 10mg at weekly intervals up to first intolerable dose (FID) or to maximum allowed dose (MAD) of 60mg/day with solifenacin 15 or 20mg/day.
  Interventions: Drug: Donepezil; Drug: Solifenacin
- Cohort 3c (Experimental): Donepezil 10mg/day upward dose titration of 5mg at weekly intervals up to first intolerable dose (FID) or to maximum allowed dose (MAD) of 40mg/day with solifenacin 15mg/day.
  Interventions: Drug: Donepezil; Drug: Solifenacin

INTERVENTIONS:
Drug: Donepezil — Donepezil dose increased at weekly intervals up to first intolerable dose (FID) or to maximum allowed dose (MAD) together with solifenacin.
Drug: Solifenacin — Donepezil dose increased at weekly intervals up to first intolerable dose (FID) or to maximum allowed dose (MAD) together with solifenacin.

SUMMARY:
This is a Phase II, ascending dose study of CPC-201 in patients with dementia of Alzheimer's type to determine the optimal dose titration schedule.

DETAILED DESCRIPTION:
This is a Phase II, ascending dose study of CPC-201 in patients with dementia of Alzheimer's type to determine the optimal dose titration schedule. The study involves a step wise cohort design in two different patient populations: Group 1 will comprise of patients who have been treated with low dose of CPC-201(5 or 10 mg/day) (given once daily) for at least 4 weeks just prior to Day1. Group 2 will consist of patients who have never been treated with CPC-201 before or who have not received any other AChEI for the past 6 months.

In this study, CPC-201 dose will be increased at weekly intervals, in accordance with the schedules given below, to its first intolerable dose (FID) or maximum allowed dose (MAD) of 60 mg/day (40mg/day for Cohort 3c) together with solifenacin 15 mg/day.

Cohort 1 1st week: 20mg 2nd week: 30mg 3rd week: 40mg 4th week: 50mg 5th week: 60mg Cohort 2* 1st week: 20mg 2nd week: 40mg 3rd week: 60mg Cohort 1b 1st - 2nd week: 10mg 3rd week: 20mg 4th week: 30mg 5th week: 40mg 6th week: 50mg 7th week: 60mg Cohort 3c* 1st week: 10mg 2nd week: 15mg 3rd week: 20mg 4th week: 25mg 5th week: 30mg 6th week: 35mg 7th week: 40mg

*: The dose titration schedule of Cohort 2 and 3 may be altered based on Cohort 1 result.

Patients will be enrolled in Cohort 2 only when patients enrolled in Cohort 1 have safely completed titration. Similary, patients will be enrolled in Cohort 3, only when patients enrolled in Cohort 2 have safely completed titration.

Patients reaching their FID or having completed one week treatment with donepezil 40mg/day, have two options.

Option 1: Patient will be allowed to immediately enter a long term extension at their Maximum tolerated dose (MTD) or MAD.

Option 2: Patients may choose not to enter the long term extension, in which case the Investigator will decide whether the patient should discontinue high dose of donepezil without down-titration, or whether donepezil should be downtitrated to their own standard of donepezil dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an Institutional Review Board (IRB) approved informed consent document
2. Aged 50 - 89 years inclusive.
3. Meeting the diagnosis of probable AD consistent with:

   * Revised National Institute on Aging-Alzheimer's Disease Association (NIA-ADA) criteria and
   * Diagnostic and Statistical Manual of Mental Disorders (DSM IV) criteria.
4. Mild to severe severity (Mini-Mental Status Exam [MMSE] scores 7 - 24 inclusive).
5. Rosen-Modified Hachinski Ischemia Score of ≤4.
6. Have a suitable caregiver to supervise the at-home administration of study drugs and observe for AEs.
7. Patients treated with donepezil 5 or 10 mg/day (given once daily) for at least 4 weeks just prior to Day1 for Population (group) 1 or;
8. Patients never been treated with donepezil before (donepezil naïve) or who have not received any other AChEI for the past 6 months for Population (group) 2.
9. Patients in generally good health as indicated by their medical history and physical examination, vital signs, electrocardiogram (ECG), and standard laboratory tests.

Exclusion Criteria:

1. Women of child bearing potential.
2. History or presence of a seizure disorder.
3. Current unstable peptic ulcer disease, urinary or gastric retention; asthma or obstructive pulmonary disease.
4. History or presence of bladder outflow obstruction, gastrointestinal obstructive disorder or reduced GI motility, or narrow-angle glaucoma.
5. History or presence of gastrointestinal, hepatic, or renal disease, or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
6. Renal and hepatic dysfunction with:

   * Total Bilirubin: >1.5 x UNL
   * AST: >2.5 x UNL
   * ALT: >2.5 x UNL
   * Serum Creatinine: >1.5 x UNL
   * Creatinine Clearance: <30 mL/min (calculated by Cockcroft and Gault equation)
7. History or presence of myasthenia.
8. History or family history of Prolonged QT Syndrome.
9. History of unexplained syncope or family history of unexplained syncope or sudden death.
10. Myocardial infarction or hospitalization for congestive heart failure within 6 months.
11. ECG findings of:

    * Complete Left Bundle Branch Block;
    * Ventricular pacing;
    * 2nd degree or 3rd degree AV block;
    * Atrial fibrillation or atrial flutter;
    * HR <45 or >100;
    * PR >220 msec; or
    * QTcF >450 msec in male, >470 msec in female
12. Known hypersensitivity to donepezil, solifenacin or related drugs.
13. History of drug significant allergy.
14. History of substance abuse, known drug addiction, or positive test for drugs of abuse or alcohol.
15. Patients treated with the following medications within 8 weeks of screening

    * AChEIs (other than donepezil),
    * Peripherally acting anticholinergics (such as drugs for the treatment of overactive bladder disorder),
    * Psychoactive medications (including antipsychotics, antidepressants, anxiolytics or sedative hypnotics) having significant anticholinergic effects and/or believed to affect cognitive function.

    Other medications are acceptable, at the investigators discretion, if dosage is held stable for at least 4 weeks prior to screening and throughout the study.
16. Patients considered unlikely to co-operate in the study, and/or poor compliance anticipated by the investigator.
17. Patients hospitalized within 4 weeks of screening.
18. Any other clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with study objectives.
19. Patients who have participated in another clinical trial with an investigational drug within previous 30 days.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn James, Study Chair — Allergan
Locations (4):
- United States (4):
  - Quantum Laboratories, Deerfield Beach, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - PMG Research, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 28 subjects between the chronological ages of 50 and 89 years with dementia of Alzheimer's type were enrolled in the study.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1b | Cohort 3c
Started | 8 | 1 | 6 | 13
Completed | 7 | 1 | 5 | 12
Not Completed | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1b | Cohort 3c | Total
Number analyzed (Participants) | 8 | 1 | 6 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72 (10.6) | 74 | 75.5 (6.9) | 73 (8.4) | 73.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 3 | 5 | 14
  Male | 2 | 1 | 3 | 8 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 1 | 5 | 11 | 25
  Black or African- American | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reached the Maximum Allowed Dose (MAD) in Their Respective Cohort
Description: Of the four cohorts with different dosing schedules for CPC-201, the cohort with the greatest proportion of participants to reach the donepezil MAD was determined to be the optimal administration regimen.
Time Frame: 1-7 weeks
Population: The MTD evaluable population was defined as all patients who completed the donepezil dose titration.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1b | Cohort 3c
Number analyzed (Participants) | 7 | 1 | 5 | 12
Participants | 2 | 0 | 1 | 6

2. Secondary Outcome: Number of Participants With TEAEs Leading to Study Drug Discontinuation
Description: Number of subjects who experienced any treatment-emergent adverse events (TEAEs) leading to study drug discontinuation
Time Frame: 1-7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1b | Cohort 3c
Number analyzed (Participants) | 8 | 1 | 6 | 13
Participants | 2 | 0 | 1 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected until week 7.
Description: All subjects who received at least one dose of any study drug.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1b | Cohort 3c
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/1 | 0/6 | 1/13
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/1 | 0/6 | 1/13
Other Adverse Events (participants affected / at risk) | 6/8 | 1/1 | 6/6 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=1) | Cohort 1b (N=6) | Cohort 3c (N=13)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=1) | Cohort 1b (N=6) | Cohort 3c (N=13)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 4 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 2
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Crying (General disorders) | 0 | 0 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Drooling (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cancer surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02549196/SAP_000.pdf
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02549196/Prot_001.pdf